CLINICAL TRIAL: NCT03275454
Title: A Phase 1 Safety, Tolerability, and Pharmacokinetics & Pharmacodynamics Study of Multiple- Dose BIVV009 in Patients With Chronic Immune Thrombocytopenia (ITP)
Brief Title: A Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple- Dose BIVV009 in Participants With Chronic Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDR16218; BIVV009-201 (Other: Bioverativ Therapeutics Inc.)
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2022-04

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: Autoimmune Diseases; Hematologic Diseases; Immune System Diseases; Blood Platelet Disorders
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Autoimmune Diseases; Hematologic Diseases; Immune System Diseases; Blood Platelet Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BIVV009 (Experimental): Participants who weigh less than 75 kilogram (kg) will receive fixed doses of 6.5 grams of BIVV009 intravenous (IV) infusion and participants who weigh 75 kg or more will receive fixed doses of 7.5 grams of BIVV009 every 2 weeks for approximately 21 weeks in Part A (based on time to complete 11 doses of study drug). There will be a 9-week safety follow-up/washout period after administration of the last dose of study drug in Part A. Participants who have been shown to benefit from BIVV009 treatment during Part A, will receive BIVV009 (based on weight) biweekly for up to 52 weeks of BIVV009 after Last Patient In (LPI) in part B.
  Interventions: Drug: BIVV009 6.5 grams; Drug: BIVV009 7.5 grams

INTERVENTIONS:
Drug: BIVV009 6.5 grams — Participants who weigh less than 75 kilogram (kg) will receive fixed doses of 6.5 grams of BIVV009.
Drug: BIVV009 7.5 grams — Participants who weigh 75 kg or more will receive fixed doses of 7.5 grams of BIVV009.

SUMMARY:
The purpose of this study is to explore the safety, preliminary clinical benefit, and activity of BIVV009 in patients with chronic immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria

Part A:

* Chronic immune thrombocytopenia (ITP) (ITP lasting for greater than or equal to ([>=] 12 months) as defined in the protocol
* Normal prothrombin time (PT/INR) and activated partial thromboplastin time (aPTT)
* No history of a coagulation disorder
* Hemoglobin level greater than (>) 10 gram per deciliter (g/dL) (following blood transfusion is acceptable) and normal white blood cell (WBC) and neutrophil counts (elevated WBC/absolute neutrophil count [ANC] attributed to steroid treatment is acceptable)
* Eastern Cooperative Oncology Group (ECOG) performance status grade less than or equal to (<=) 2
* Documented vaccinations against encapsulated bacterial pathogens (Neisseria meningitis, including serogroup B meningococcus [where available], Haemophilus influenzae, and Streptococcus pneumoniae) within 5 years of enrollment
* Adequate intravenous (IV) access

Part B:

* Able to comprehend and to give informed consent for Part B
* History of ITP and previously treated with at least 1 dose of BIVV009 in Part A
* Evidence of treatment efficacy to BIVV009 as defined by a platelet count > 30*10^9/L on at least 1 occasion OR a doubling of the platelet count from baseline
* Participants who have completed the 21-week Part A treatment period but have not reached the Part A End of Study (EOS) visit must have evidence of ongoing or recurrent thrombocytopenia during the Part A safety follow-up/washout period as demonstrated by a platelet count less than (<) 50*10^9/L or a >= 50 percent (%) decrease in platelet count over < 1 week

Exclusion Criteria:

Part A:

* Clinically significant medical history or ongoing chronic illness that would jeopardize the safety of the participant or compromise the quality of the data derived from his/her participation in this study
* Clinically relevant infection of any kind within the preceding month of enrollment
* History of venous or arterial thrombosis within the preceding year of enrollment
* Use of aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), or anticoagulants within 1 week of enrollment
* Clinical diagnosis of systemic lupus erythematosus (SLE) or other active autoimmune disorders associated with anti-nuclear antibodies (ANAs) including those that are medically controlled, at Screening (other than ITP)
* Secondary immune thrombocytopenia from any cause including lymphoma, chronic lymphocytic leukemia, and drug-induced thrombocytopenia
* Positive hepatitis panel (including hepatitis B surface antigen and/or hepatitis C virus antibody) prior to or at Screening
* Positive human immunodeficiency virus (HIV) test result prior to or at Screening

Part B:

* Presence of unacceptable side effects or toxicity associated with BIVV009 (including prior hypersensitivity reactions to BIVV009) such that there is an unfavorable risk-benefit assessment for continued treatment with BIVV009 in the opinion of the Investigator and/or Sponsor
* For participants who have completed the 9-week safety follow-up/washout period and final study visit before entry into Part B, a positive hepatitis panel (including hepatitis B surface antigen and/or hepatitis C virus antibody) prior to or at Screening. Patients who have undergone hepatitis C antiviral therapy may be allowed if they are documented to be negative for hepatitis C virus ribonucleic acid (RNA) on at least 2 occasions separated by at least 3 months (including 1 RNA test at least 6 months after completion of antiviral therapy) and are also negative for hepatitis C virus RNA at Screening
* Use of prescribed or over-the-counter medications, supplements, vitamins, and/or herbal remedies within 2 weeks before the first dose of BIVV009 in Part B, which in the judgment of the Investigator may adversely affect the participants welfare or the integrity of the study results (excluding hormonal contraception in female participants)
* If previously treated with rituximab, the last dose of rituximab was administered < 12 weeks before the first dose of BIVV009 in Part B
* Clinical diagnosis of systemic lupus erythematosus (SLE) or other active autoimmune disorders associated with anti-nuclear antibodies (ANA), including those that are medically controlled, at Screening (other than ITP). Positive ANAs at screening that are not associated with an autoimmune disorder (other than ITP) may be allowed if present for >= 28 days without associated clinically relevant symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 97 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. A serious adverse event (SAE) is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Number of Participants With Premature Study Terminations | Approximately 97 weeks
  Number of participants with premature study terminations will be assessed.
Number of Participants With Clinical Laboratory Abnormalities | Approximately 97 weeks
  Clinical laboratory abnormalities including one or more specific target-organs for toxicity of BIVV009, abnormalities in D-dimer, thrombin-anti-thrombin assay, and Systemic Lupus Erythematosus (SLE) panel.

SECONDARY OUTCOMES:
Part A: Change From Baseline in Peripheral Blood Platelet Count at Part A End of Treatment (A-EOT) | Baseline and A-EOT (Day 147)
  Change from baseline in peripheral blood platelet count at A-EOT will be assessed.
Part A: Change From Baseline in Peripheral Blood Platelet Count during BIVV009 Treatment | Baseline up to Day 147
  Change from baseline in peripheral blood platelet count during BIVV009 treatment will be assessed.
Part A: Number of Participants who are independent from using combination Immune Thrombocytopenia (ITP) therapy during A-EOT but receive combination ITP therapy after A-EOT | Day 147 (A-EOT) up to Day 196 (EOS)
  Number of participants who are independent from using combination ITP therapy during A-EOT but receive combination ITP therapy after A-EOT will be assessed.
Part A: Number of Participants who Achieve Complete Response Through A-EOT | Up to Day 147
  Complete response (CR) is defined as a platelet count greater than or equal to (>=) 100*10^9/liter (L) measured on 2 occasions at least 7 days apart and the absence of bleeding on and through these two visits and the lack of combination ITP therapy on and through these two visits.
Part A: Number of Participants who Achieve Response Through A-EOT | Up to Day 147
  Response or Better: Response (R) is defined as a platelet count >= 30*10^9/L and a greater than 2-fold increase from baseline measured on 2 occasions at least 7 days apart and the absence of bleeding on and through these two visits and the lack of combination ITP therapy on and through these two visits; and CR: A platelet count >=100*10^9/L measured on 2 occasions at least 7 days apart and the absence of bleeding on and through these two visits and the lack of combination ITP therapy on and through these two visits.
Part A: Duration of Complete Response per Each CR | Up to Day 196
  Duration of CR is defined as the number of consecutive days in which a patient's peripheral blood platelet count is >= 100*10^9/L and the absence of bleeding, and the lack of platelet transfusions or other ITP therapy.
Part A: Duration of Response per Each Response | Up to Day 196
  Duration of response is defined as the number of consecutive days in which a patient's peripheral blood platelet count is >= 30*10^9/L and the absence of bleeding, and the lack of platelet transfusions or other ITP therapy.
Part A: Time to First Platelet Response | Up to Day 196
  Time to first platelet response is defined as greater than or equal to 30*10^9/L, 50*10^9/L, 100*10^9/L (confirmed by a consecutive platelet response at least 7 days apart).
Part A: Number of Participants who Report Loss of Response Among Those who Achieve Response | Up to Day 196
  Number of participants who report loss of response among those who achieve response will be reported. For a participant with a response (R), the loss of the response is defined as a platelet count < 30*10^9/L measured on 2 consecutive occasions at least 1 day apart, or a less than 2-fold increase in platelet count from baseline measured on 2 consecutive occasions at least 1 day apart, or the presence of bleeding, or use of the combination ITP therapy.
Part A: Number of Participants who Report Loss of Complete Response Among Those who Achieve Complete Response | Up to Day 196
  Number of participants who report loss of complete response among those who achieve complete response will be reported. For a participant with a complete response (CR), loss of complete response is defined as a platelet count less than (<) 100*10^9/L measured on 2 consecutive occasions more than 1 day apart and/or the presence of bleeding or use of the combination ITP therapy.
Part B: Change From Baseline in Peripheral Blood Platelet Count to B-EOT | Baseline up to 52 weeks
  Change from baseline (Part B) in peripheral blood platelet count to B-EOT will be assessed.
Part B: Number of Participants who Achieve CR and the Lack of Platelet Transfusions or Other ITP Therapy During Treatment Period | Up to 52 weeks
  Number of participants who achieve CR and the lack of platelet transfusions or other ITP therapy during Part B treatment period will be reported. Complete response (CR): A platelet count >= 100*10^9/L measured on 2 occasions at least 7 days apart and the absence of bleeding on and through these two visits and the lack of combination ITP therapy on and through these two visits.
Part B: Number of Participants who Achieve Response Through Part B End of Treatment (B-EOT) | Up to 52 weeks
  Number of participants who achieve response through B-EOT will be reported.
Part B: Duration of Complete Response per Each CR | Up to 52 weeks
  Duration of CR is defined as the number of consecutive days in which a participant's peripheral blood platelet count is >= 100*10^9/L and the absence of bleeding, and the lack of platelet transfusions or other ITP therapy.
Part B: Duration of Response per each Response | Up to 52 weeks
  Duration of response is defined as the number of consecutive days in which a participant's peripheral blood platelet count is >= 30*10^9/L and the absence of bleeding, and the lack of platelet transfusions or other ITP therapy.
Part B: Number of Participants who achieve a platelet count >= 100*10^9/L on 2 consecutive occasions at least 7 days apart and have the absence of bleeding on and through these two visits and use any combination ITP therapy through B-EOT | Up to 52 weeks
  Number of participants who achieve a platelet count >= 100*10^9/L on 2 consecutive occasions at least 7 days apart and have the absence of bleeding on and through these two visits and use any combination ITP therapy through B-EOT will be assessed.
Part B: Number of Participants who achieve a platelet count >=30*10^9/L, a >2-fold increase from baseline measured on 2 consecutive occasions at least 7 days apart, have absence of bleeding on and through these two visits, use any combination ITP therapy | Up to 52 weeks
  Number of participants who achieve a platelet count >= 30*10^9/L and a greater than (>) 2-fold increase from baseline measured on 2 consecutive occasions at least 7 days apart and have the absence of bleeding on and through these two visits and use any combination ITP therapy through B-EOT will be assessed.
Part B: Number of Participants who do not Require Other Immune Thrombocytopenia (ITP) Therapy (non-transfusion) During the Part B Treatment Period | Up to 52 weeks
  Number of Participants who do not require other ITP therapy (non-transfusion) following the last BIVV009 dose will be assessed.
Part B: Number of Participants who do not Require Platelet Transfusions During the Part B Treatment Period | Up to 52 weeks
  Number of Participants who do not require platelet transfusions during the Part B treatment period will be reported.
Part B: Number of Participants who Experience any Bleeding Episode, Bleeding by Grade or Serious Bleeding | Up to 52 weeks
  Number of participants who experience any bleeding episode, bleeding by grade or serious bleeding according to the International Working Group (IWG) Bleeding Assessment Tool (BAT) will be reported.
Plasma Concentrations of BIVV009 | Approximately 97 weeks
  Plasma concentrations of BIVV009 will be assessed.
Maximum Observed Plasma Concentration (Cmax) of BIVV009 | Approximately 97 weeks
  Maximum observed concentration of BIVV009 in plasma will be assessed.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of BIVV009 | Approximately 97 weeks
  Time to Reach Maximum Observed Plasma Concentration (Tmax) of BIVV009 will be assessed.
Area Under the Concentration-time Curve (AUC) From Hour 0 to the last quantifiable time point (AUC [0-t]) of BIVV009 | Approximately 97 weeks
  AUC (0-t) is the area under the Concentration-time curve (AUC) from hour 0 to the last quantifiable time point of BIVV009.
Number of Participants With Anti-drug antibodies (ADAs) Against BIVV009 | Up to 97 weeks
  Blood samples will be collected to determine number of participants with anti-drug antibodies (ADAs) against BIVV009.
Complement System Classical Pathway Levels as Measured by WIESLAB Assay | Up to 97 weeks
  Inhibition by BIVV009 of the complement system classical pathway measured by the WIESLAB assay.
Total Complement (CH50) Levels | Up to 97 weeks
  Complement CH50 is a blood test that helps us determine whether protein abnormalities and deficiencies in the complement system are responsible for any increase in autoimmune activity. It will be assessed using complement assays.
Total Complement Factor C4 Levels | Up to 97 weeks
  Total C4 Levels will be assessed in plasma using complement assays.
C1 Complex Components: C1q | Up to 97 weeks
  C1q Levels will be assessed in plasma using complement assays.
Thrombopoietin Level | Up to 97 weeks
  Thrombopoietin level will be assessed in plasma using complement assays.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- United States (3):
  - Georgetown Lombardi Comprehensive Cancer Center, Georgetown, District of Columbia
  - Massachusetts General Hospital - Cancer Center, Boston, Massachusetts
  - University of Pittsburgh Medical Center (UPMC) Hilman Cancer Center, Pittsburgh, Pennsylvania
- Essen University Hospital Department of Hematology, Essen, Germany
- University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Broome CM, Roth A, Kuter DJ, Scully M, Smith R, Wang J, Reuter C, Hobbs W, Daak A. Safety and efficacy of classical complement pathway inhibition with sutimlimab in chronic immune thrombocytopenia. Blood Adv. 2023 Mar 28;7(6):987-996. doi: 10.1182/bloodadvances.2021006864. PMID 35973190